CLINICAL TRIAL: NCT03343574
Title: Exercise and Its Cardiovascular Effects in Patients of Parkinson's Disease With Cardiovascular Autonomic Dysfunction
Brief Title: Cardiovascular Effects of Exercise in Patients With Parkinson's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faizan Ahmed (Other)
Responsible Party: Sponsor-Investigator, Faizan Ahmed, Study coordinator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSREB109386
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease; Orthostatic Hypotension
Keywords: Parkinson's Disease; Neurogenic orthostatic hypotension; Orthostatic intolerance; Exercise; Abdominal binder; Autonomic dysfunction; Dizziness; Physical Therapy; Blood pressure; Heart rate; Autonomic function testing; Neurology; Falls risk; Autonomic Nervous System; Autonomic reflex screening; Cerebral blood flow; Cerebral perfusion; Activities of Daily Living
MeSH Terms: conditions — Parkinson Disease; Hypotension, Orthostatic; Orthostatic Intolerance; Motor Activity; Primary Dysautonomias; Dizziness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal Strengthening Exercise (Experimental): All participants in this arm shall perform exercises for the strengthening of abdominal muscles for a period of three months in addition to the routine care provided to them for the management of Parkinson's Disease. The exercises are structured and need to be performed on a routine basis.
  Interventions: Other: Abdominal Strengthening Exercise
- Routine Care (No Intervention): All participants in this group shall continue to obtain routine care for the management of Parkinson's Disease.

INTERVENTIONS:
Other: Abdominal Strengthening Exercise — Abdominal strengthening exercises involve the muscles of the abdomen. These exercises are to be done in different positions like lying down (recumbent) position, sitting and standing positions. The person performing the exercise contracts the abdominal muscles for a predetermined number of times (up to 10 times), holds the contracted position for up to 10 seconds and then releases the contraction to relax and return to the original state. These exercises are done for three times everyday.
  Other Names: Abdominal Exercise
  Arms: Abdominal Strengthening Exercise

SUMMARY:
Abnormalities in the regulation of cardiovascular system due to autonomic nervous system (ANS) dysfunction may lead to a sudden decline in blood pressure (BP) upon standing, sitting or performing activities/exercises in patients with Parkinson's Disease (PD). This sudden decline in BP is known as 'orthostatic hypotension' (OH). OH may cause dizziness and/or black-outs, which may increase the risk of falls. As falls are potentially dangerous and disabling, it is important to prevent their occurrence. Keeping BP within normal range upon change of posture or with activities is therefore of great significance. Pooling of blood in the abdominal blood vessels may be one of the reasons for OH to happen. This research focuses on strengthening the weak abdominal muscles of the participants so that the compressive action of these muscles can help decrease such pooling. Therefore, the researchers hypothesize that strengthening the abdominal muscles shall prove to be helpful in controlling orthostatic hypotension by preventing a sudden decline in blood pressure of the participants upon assumption of upright posture. The secondary hypothesis is that there exists a significant difference in the response of the cardiovascular system to a variety of postures/activities/exercises when patients of PD having cardiovascular autonomic dysfunction are compared with patients of PD with normal ANS function.

This study has two parts - stage 1 and stage 2. Only stage 2 is a randomized controlled trial. Stage 1 involves testing the functional integrity of the autonomic nervous system, and observation of the cardiovascular responses of the participants to different postures/activities/exercises and to the use of an abdominal binder (which is a compressive garment worn around the abdomen). Findings of stage 1 shall help the researchers better understand the cardiovascular abnormalities present in such patients at rest and with activity. Stage 2 involves strength training for the abdominal muscles that is to be done by the participant at her/his residence for a period of 3 months followed by a second round of autonomic function testing and observation of the cardiovascular responses to the use of abdominal binder. Findings of stage 2 shall help the researchers determine if strength training of the abdominal muscles can be a useful strategy to counter the cardiovascular abnormalities found in the participants during the testing in stage 1.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is associated with abnormal control of the cardiovascular system in up to 50% of patients. The cardiovascular autonomic dysfunction is a result of abnormal regulation of the cardiovascular system by the autonomic nervous system (ANS). It manifests as orthostatic hypotension, supine hypertension, and may possibly involve abnormal heart rate and rhythm, as well as abnormal haemodynamic responses to exercise. Orthostatic hypotension is a sudden decline in the blood pressure (BP) as a result of assumption of more upright posture like standing up and may present as a generalized weakness, light-headedness, mental "clouding" up to syncope. Moreover, the stress of exercise may worsen the manifestation of an asymptomatic cardiovascular autonomic dysfunction, resulting in decreased balance control which may render the patient unable to exercise and/or predispose the patient to a higher risk of falls, decreased ability in activities of daily living (ADLs) and confusion. Falls in elderly patients, which constitute the majority of patients with PD, are potentially dangerous and disabling. However, the response of the cardiovascular system to neither the routinely prescribed physiotherapeutic exercises nor the routine physical activities of the patients of PD are known. Thus, due to lack of any research data on the effects of these exercises/activities it cannot be determined whether certain components of the routine physiotherapy treatment are appropriate and safe for the patient with regard to the development or worsening of cardiovascular autonomic dysfunction. The same is true for some of the patient's ADLs that may trigger signs and symptoms of cardiovascular autonomic dysfunction. The researchers, therefore, intend to investigate the same.

This research has two parts - stage 1 and stage 2. Only stage 2 is a randomized controlled trial. The specific objectives pertaining to each stage are:

Stage 1 - To analyze the spectrum of cardiovascular dysfunction in patients with PD -

* As determined by the autonomic reflex screening; and
* In response to the different postures/activities/exercises and to wearing an abdominal binder.

Stage 2 - To investigate whether strengthening of the abdominal muscles can be an effective strategy to improve cardiovascular system's ability to counter the development of OH.

Stage 1:

Upon inclusion into the study, baseline autonomic reflex screening shall be undertaken. This screening has the following components:

1. Quantitative Sudomotor Axon Reflex Test (QSART): The QSART evaluates the postganglionic sympathetic sudomotor axon i.e. it evaluates the response of the sweat cells which are controlled by the ANS to acetylcholine (ACh). For this, participant's skin is cleaned and prepared at four sites. Then, ACh is applied at those sites. The movement of ACh across the skin is facilitated by iontophoresis (using low intensity electrical current of 2 mA).

   Recordings are made for 5 minutes with stimulus application followed by an additional 5 minutes after stimulus termination.

   For the subsequent 3 tests in the autonomic reflex testing, participants are instrumented with a beat-to-beat blood pressure device and three-lead electrocardiogram (ECG).
2. Heart Rate Response to Deep Breathing (HRDB) with the participant supine: A 1-minute baseline is recorded. Immediately thereafter, eight consecutive breathing cycles will take place. Each breathing cycle consists of maximal inspiratory and expiratory phases of 5 seconds each. Visual feedback is provided to ensure breathing consistency. The procedure is repeated after a 2-minute rest period.
3. Beat-to-beat BP response to Valsalva Maneuver: The participant, in the supine position is asked to exhale after a deep inhalation while maintaining a column of mercury at 40 mm for 15 seconds while blowing the air out via a tubing with an air leak. The maneuver is repeated until two similar beat-to-beat BP and HR are attained. Each maneuver is separated by 3-minute rest.
4. Head-up Tilt: The participant is secured to an automated tilt-table. A 5-minute recording of HR and BP is obtained while the patient is supine. The table is tilted slowly to 70 degrees over the course of 10 seconds (it is similar to standing up). Subjects remain tilted for 5 minutes or until one of the stopping criterion is met. Manual BP in addition to automated BP may be taken 1 minute before the tilt, at 1, 3, and 5 minutes during head tilt-up and 1-minute post head tilt-up. All automated parameters are displayed on a computer console. The specific stopping rules are 1) patient request, 2) presyncope, and 3) rapid decline in systolic blood pressure in response to tilt. If any of these are met, the patient will be placed back into supine position.

The five primary endpoints of autonomic reflex testing are:

1. total sweat volume on QSART;
2. HR variation on HRDB;
3. Valsalva ratio during the Valsalva maneuver;
4. HR change in response to head-up tilt; and
5. BP change in response to head-up tilt. The severity and distribution of the autonomic dysfunction will be quantified using the Composite Autonomic Severity Score (CASS).

Blood flow velocity in the Middle Cerebral Artery (MCA) and frontal/prefrontal cortical perfusion will be measured using Trans-Cranial Doppler (TCD) and functional Near-Infrared Spectroscopy (fNIRS). For TCD, a Velcro head band with a flat probe will be placed on the subject's head before any autonomic test is done and blood flow velocities will be recorded before any autonomic testing for 5 minutes. After TCD is finalized, fNIRS will be acquired while the patient performs each maneuver in the rest of the protocol. The participant will be lying down with the fNIRS probes (two emission and four detection) positioned on the forehead. The probes are held securely in position by a holder that includes a Velcro strap wrap around the head. This probe location will provide sensitivity to the prefrontal cortex, which is known to be activated by information processing tasks. For the following maneuvers in the rest of the protocol, the fNIRS probes will be placed at the C3 location (i.e., above the primary motor cortex) according to the international 10-20 system for EEG electrode placement. fNIRS is a non-invasive optical method that can be used to detect cortical activity at the bedside. fNIRS systems use the wave length-dependent absorption property of hemoglobin to monitor changes in the brain concentration of oxy- and deoxyhemoglobin during a functional task [analogous to functional MRI (fMRI)]. The ratio between oxy- and deoxyhemoglobin allows estimating cortical perfusion. fNIRS data will complement the TCD information. TCD provides information regarding MCA flow velocity, allowing us to estimate pial arteries flow velocities, while fNIRS provides information regarding changes in cortical perfusion, and thus, intraparenchymal arteries vasoconstriction.

After this, we shall record a six-month retrospective history of falls. Dizziness Handicap Inventory (DHI), Autonomic Symptom Profile (ASP), University of California Los Angeles Dizziness Questionnaire (UCLA-DQ), Orthostatic Hypotension Questionnaire (OHQ) and the Orthostatic Discriminant and Severity Scale (ODSS) shall be used to assess and quantify the influence of autonomic dysfunction, orthostatic hypotension and dizziness on participant's life.

After the above mentioned baseline evaluation of the participant is over, the participant shall be tested for cardiovascular responses to different postures/activities/exercises and to the use of an abdominal binder. For this, the participants shall be required to undergo recording of BP, heart rate (using ECG), analysis of blood flow velocity in the MCA and frontal/prefrontal cortical perfusion (as described above) while performing any/some of the following exercises in any sequence or combination:

* Deep breathing exercise while in sitting position in a chair or in a standing position, with or without breath-hold;
* Sit-to-stand from a chair and return stand-to-sit into the same chair;
* Shoulder elevation and/or elbow flexion-extension exercise while holding a 500 ml water bottle (filled) in each hand (in standing position);
* Tandem walking (to walk on a straight line where the toes of the back foot touch the heel of the front foot at each step);
* Single leg standing (for each leg);
* Cross-legged standing;
* Supine cycling exercise;
* Stationary bicycle exercise;
* Abdominal muscle contraction exercise; and
* Compression of the abdomen using an abdominal binder. An abdominal binder is a fitted elastic garment that is used for compression of the abdominal wall. It is available in different sizes. It can be used to support the muscles of the abdominal wall.

The participants will undergo supine/stationary bicycle exercise for a maximum of 12 minutes in order to produce sympathetic ANS activation. The stationary bicycle will be adapted based on the limitations of the individual at a steady workload. Maximum safe workload will be calculated using Karvonen/Heart Rate Reserve formula, according to the current guidelines. After a 1-min warm-up period at a 0 Watts workload, an exercise load of 10 Watts/min will be added and maintained for the full 12 minutes, unless an aspect of the stopping criteria is met. The specific stopping rules are 1) patient request, 2) rapid decline in systolic blood pressure, and 3) researcher/staff member's decision to terminate the exercise for participant's safety.

All participants shall be required to complete stage 1. However, only those participants who have significant autonomic dysfunction shall proceed to stage 2 of the study.

Stage 2:

Patients identified with autonomic dysfunction using the autonomic reflex screening (in stage 1) shall be randomly allocated to either of the two groups. The groups shall be labelled as group 'Abdominal strengthening exercises' (experimental) and group 'Routine care' (control). Patients in the experimental group shall in addition to the routine care perform abdominal strengthening exercises for three months at their home and maintain an exercise log sheet, whereas, patients in the control group shall continue with the routine care for the next three months. During the follow-up at three months, patients in both the groups will again undergo the same testing as mentioned in stage 1.

Abdominal strengthening exercises involve the muscles of the abdomen. Abdominal muscles are contracted after the participant assumes different postures for a predetermined duration and for a predetermined number of times in a day. The two groups shall be compared for effectiveness of abdominal strengthening exercises in preventing orthostatic hypotension upon autonomic reflex testing after 3 months. Both groups shall additionally be compared while wearing abdominal binder during a second tilt testing. A three-month history of falls will be recorded and all participants shall be asked to answer the four questionnaires i.e. DHI, ASP, OHQ and ODSS again.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's Disease;
* Between stages 2 and 4 of Hoehn and Yahr classification of Parkinson's Disease;
* Male or female; and
* Age 40-90 years.

Exclusion Criteria:

* Therapy with anticholinergic, alpha- and beta-adrenergic antagonists or other medication, which could interfere with the regulation of blood pressure and heart rate. These medications are commonly used to treat conditions such as irregular heartbeats, high blood pressure, heart failure, urinary incontinence and other medical conditions (e.g. Alprazolam (Xanax), Amantadine (Symmetrel), Baclofen, Cimetidine, Codeine. Doxazosin, Prazosin, Atenolol (Tenormin), Bisoprolol (Zebeta, also sold as Ziac), Carvedilol (Coreg), Propranolol (Inderal, Inderal LA);
* Clinically significant coronary artery disease;
* Presence of nerve damage in the peripheral nervous system;
* Pregnant or breast feeding females; and
* The presence of failure of other organ systems or diseases that can affect autonomic function or the participant's ability to cooperate. These include dementia, specific tumors, heart failure, hypertension, renal or hepatic disease, severe anemia, alcoholism, hypothyroidism, surgical procedures where the nerves of the sympathetic nervous system have been cut, or cerebrovascular disease.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2024-11-28 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | up to 3 hours for each visit. A total of 2 visits are expected for each participant.
  Continuous non-invasive monitoring using a finger cuff. Blood Pressure will be measured in millimetres of Mercury (mmHg).

SECONDARY OUTCOMES:
Heart Rate | up to 3 hours for each visit. A total of 2 visits are expected for each participant.
  Continuous non-invasive monitoring of rate and rhythm of the beating of the heart. It will be measured in beats per minute.
Composite Autonomic Severity Score | Up to one hour for autonomic reflex testing for each visit. A total of 2 visits are expected for each participant.
  This score is the result of the autonomic reflex testing. It combines the sweat volume (in micro-litres), heart rate and blood pressure findings from the autonomic reflex test to provide a discrete numerical value.
Middle Cerebral Artery flow velocity | Up to three hours for each visit. A total of 2 visits are expected for each participant.
  Continuous monitoring and periodical recording of blood flow velocity in the Middle Cerebral Artery of the brain. It is based on ultrasound technology and is measured on both sides of the head of the participant (left and right sides). The blood flow velocity is expressed in centimetres per second.
Changes in the ratio between oxy- and deoxy-hemoglobin | Up to three hours for each visit. A total of 2 visits are expected for each participant.
  This score is obtained using the Functional Near-Infrared Spectroscopy. This is expressed as a numerical value which has no unit of measurement.
The Composite Autonomic Symptom Scale (COMPASS) | 20 minutes
  The Autonomic Symptom Profile Questionnaire uses the COMPASS scale to generates a score that is obtained using the Autonomic Symptom Profile questionnaire (which is a paper-based self-completed (complete by the patient) questionnaire containing 169 items). The results are expressed in numerical values. The questionnaire evaluates 10 domains related to the functioning of the autonomic nervous system. Higher scores indicate more or worse symptoms. The maximum score for men can be 200 and for women it can be 170, in addition to the 12 questions pertaining to psychosomatic problems where each question carries a maximum score of 10. The autonomic symptom profile questionnaire is used to determine the severity of the symptoms of autonomic nervous system dysfunction.
Orthostatic Discriminant and Severity Scores | 10 minutes
  These scores are obtained using the Orthostatic Discriminant and Severity Scale (ODSS). They are expressed in numerical values. ODSS scale will be used to quantify and discriminate orthostatic symptoms (i.e. symptoms manifested due to low blood pressure upon standing up) from non-orthostatic symptoms (i.e. symptoms which are not caused by low blood pressure upon standing up). ODSS questionnaire is a self-completed instrument and contains 33 questions. There are two types of questions - those that target orthostatic symptoms and others that target non-orthostatic symptoms, thus generating a numerical 'orthostatic score' and a numerical 'non-orthostatic score', respectively. The maximum and minimum orthostatic scores can be 107 and 7, respectively. The maximum and minimum non-orthostatic scores can be 72 and 7, respectively. Higher scores indicate more or worse affected condition of the research participant.
Orthostatic Hypotension Questionnaire Score | 5 minutes
  This score is obtained using the Orthostatic Hypotension Questionnaire. It is expressed in numerical values. The maximum score can be 100 and the minimum score can be zero. This questionnaire is self-completed by the research participant and it is used to determine how low blood pressure symptoms affect the research participants daily life. Higher scores indicate more or worse affected condition of the research participant.
Dizziness Handicap Inventory score | 5 minutes
  This score is obtained using the Dizziness Handicap Inventory. It is expressed in numerical values. The Dizziness Handicap Inventory is a self-completed instrument designed to determine the difficulties the research participant may be facing because of his/her problem of dizziness. It has two parts. The first part has 25 questions divided into 3 domains. The maximum score for part 1 can be 100 and the minimum score can be zero. Part 2 of this instrument has one question with six possible answers. The maximum score for part 2 can 5 and the minimum score can be zero. Higher scores indicate that the research participant is facing greater difficulties in his/her daily life due to the presence of dizziness.

CONTACTS AND LOCATIONS:
Overall Officials: Mandar Jog, MD, Principal Investigator — Western University, London, ON
Locations (1):
- University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dubow JS. Autonomic dysfunction in Parkinson's disease. Dis Mon. 2007 May;53(5):265-74. doi: 10.1016/j.disamonth.2007.02.004. No abstract available. PMID 17656188
- [Background] Ziemssen T, Reichmann H. Cardiovascular autonomic dysfunction in Parkinson's disease. J Neurol Sci. 2010 Feb 15;289(1-2):74-80. doi: 10.1016/j.jns.2009.08.031. Epub 2009 Sep 8. PMID 19740484
- [Background] Diop M, St Lawrence K. Improving the depth sensitivity of time-resolved measurements by extracting the distribution of times-of-flight. Biomed Opt Express. 2013 Mar 1;4(3):447-59. doi: 10.1364/BOE.4.000447. Epub 2013 Feb 15. PMID 23504445
- [Background] Karvonen J, Vuorimaa T. Heart rate and exercise intensity during sports activities. Practical application. Sports Med. 1988 May;5(5):303-11. doi: 10.2165/00007256-198805050-00002. PMID 3387734
- [Background] Pina IL, Balady GJ, Hanson P, Labovitz AJ, Madonna DW, Myers J. Guidelines for clinical exercise testing laboratories. A statement for healthcare professionals from the Committee on Exercise and Cardiac Rehabilitation, American Heart Association. Circulation. 1995 Feb 1;91(3):912-21. doi: 10.1161/01.cir.91.3.912. No abstract available. PMID 7828326
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886